CLINICAL TRIAL: NCT05699005
Title: Comparison of an Individualized Transfusion Strategy to a Conventional Strategy in Patients Undergoing Peripheral Veno-arterial ECMO for Refractory Cardiogenic Shock: a Randomized Controlled Trial - ICONE
Brief Title: Individualized or Conventional Transfusion Strategies During Peripheral VA-ECMO
Acronym: ICONE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Amiens University Hospital (Other); University Hospital, Caen (Other); University Hospital, Rouen (Other); Centre Hospitalier Universitaire Dijon (Other); Centre hospitalier de Dunkerque (Unknown); Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020_04; 2021-A01925-36 (Other: ID-RCB number, ANSM); PHRCI-19-032 (Other: AAP number, DGOS)
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-01

CONDITIONS: Cardiogenic Shock; Extracorporeal Membrane Oxygenation; Transfusion Related Complication; Anemia; Oxygen Delivery
Keywords: ECMO; ECLS; Refractory cardiogenic shock; Transfusion; ScVO2; Outcome
MeSH Terms: conditions — Shock, Cardiogenic; Anemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and datamanagement responsible for statistical analysis will be blinded of the patient allocation group until the study completion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individulised transfusion strategy group (Experimental): Patients will recieve red blood cells transfusion in case of a drop of ScVO2 <65% after an assessment for the optimisation of SaO2 normalisation (SaO2>94%), volume optimisation, ECMO output increase, Fever (body temperature 38°3 C°), Anxiety and Pain
  Interventions: Drug: Packed Red Blood Cells (PRBCs)
- Conventionnal transfusion strategy group (Active Comparator): Transfusion will be performed in case of a hemoglobin drop <9 g/dL
  Interventions: Drug: Packed Red Blood Cells (PRBCs)

INTERVENTIONS:
Drug: Packed Red Blood Cells (PRBCs) — Patient will recieve PRBCs transfusion only in case of ScVO2 level<65% after assessment of patient for optimisation of SaO2 targeting 100%, volume status, ECMO flow (increase to 20% in relevant), pain, anxiety and fever (body temperature >38°3).
  In both groups transfusion may be performed in case massive bleeding according to local protocols, STEMI, Hyperlactatemia >4 that can be related to oxygen demand and supply DO2/VO2 ratio impairement, in all groups, transfusion should be performed in case of hemolobin level <7g/dL or worsening of neurological condition (Increase in Neurological SOFA component of 1 and more) related to DO2/VO2 impairement.
  Other Names: ScVO2 assesment to guide transfusion

SUMMARY:
This multicenter randomized controlled trial compare two transfusion strategies of red blood cells transfusion in patients supported by veno-arterial extracorporeal membrane oxygenation for refractory cardiogenic shock.

An individualized transfusion strategy based on ScVO2 level, is compared to a conventionnal strategy based on predefined hemoglobin threshold. The primary endpoint is the consumption of packed red blod cells, secondary endpoints are subgroup analysis, mortality, morbidity, and cost-effectiveness

DETAILED DESCRIPTION:
Peripheral VA-ECMO is the mainstay of mechanical circulatory support in refractory cardiogenic shock. This treatment is associated with a high consumption of packed red blood cells (PRBCs), which can reach 1 to 3 units of PRBCs per day of support. The main reasons for such a high consumption of PRBCs are the very frequent hemorrhagic complications and the prevalence of anemias not directly related to the hemorrhagic episodes. These anemias are frequent during VA-ECMO support owing to hemolysis, hemodilution, previous bleeding episodes, thrombosis, etc.

In order to restore, maintain, or increase oxygen delivery (DO2) to peripheral organs, RGCs are often performed when anemia is observed. Several studies have reported an association between transfusion of these PRBCs with morbidity and mortality in this ECMO setting.

There is no appropriate strategy to reduce PRBC consumption, taking into account other determinants of DO2. In addition, there is currently no validated or consensus hemoglobin threshold to guide transfusion in this specific population. Furthermore, this predefined threshold-based approach may be inappropriate in the setting of VA-ECMO due to differences in DO2 requirements between patients based on their etiology, disease severity, and ECMO modality. In addition, large variations in DO2 can be observed in the same patient and between ECMO settings. Therefore, a more individualized strategy guided by a DO2 surrogate, ScVO2, may be more appropriate in this population. This ScVO2 approach has recently been shown to be associated with reduced PRBCs in two randomized controlled trials in cardiac surgery patients.

The objective of this multicenter randomized controlled trial is to compare two red cell transfusion strategies in patients receiving extracorporeal veno-arterial membrane oxygenation for refractory cardiogenic shock.

An individualized transfusion strategy based on ScVO2 level is compared with a conventional strategy based on a predefined hemoglobin threshold. The primary endpoint is red blood cell consumption, the secondary endpoints are subgroup analysis, mortality, morbidity, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and older,
* supported by peripheral VA-ECMO
* for cardiogenic shock
* Life expentency >90 days
* Central venous line available ScVO2 measurement

Exclusion Criteria:

* Pregnancy,
* Lack of health insurance,
* Opposition to blood transfusion,
* Known congenital hemoglobin disease or disorder,
* Metabolic alcaloosis with pH>7.8,
* eCPR,
* Legally incapacitated adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Number of PRBCs transfused per VA-ECMO day of support | From randomisation until VA-ECMO weanning assessed up to 28 days
  Total number of PRBCs transfused during support adjusted for VA- ECMO duration

SECONDARY OUTCOMES:
Number of PRBCs transfused per VA-ECMO day of support in postcardiotomy patients | From randomisation until VA-ECMO weanning assessed up to 28 days
  Total number of PRBCs transfused during support adjusted for VA- ECMO duration in patients that underwent cardiac surgery
Total number of PRBCs transfused during the 28-day following cannulation | From randomisation until 28 days
  Total number of PRBCs transfused during the 28-day following cannulation
Changes in hemoglobin levels during VA-ECMO support | From randomisation until VA-ECMO weanning assessed up to 28 days
  daily hemoglobin levels
Changes in ScVO2 levels during VA-ECMO support | From randomisation until VA-ECMO weanning assessed up to 28 days
  daily ScVO2 levels
Changes in vosoactive index score levels during VA-ECMO support | From randomisation until VA-ECMO weanning assessed up to 28 days
  daily vasoactive index score levels
Mortality under ECMO support | From randomisation until VA-ECMO weanning assessed up to 28 days
  All cause mortality before ECMO weaning
90-day Mortality | 90 days from cannulation
  All cause mortality from cannulation untill 90 days
ECMO removal modalities | From randomisation until VA-ECMO weanning assessed up to 28 days
  Proportion of patients that according to each reason for removal ( Recovery, heart transplantation, Left ventricle or biventricle assist device or death under support)
Duration of mechanical ventilation | 28 days from cannulation
  Duration of mechnanical ventilation from cannulation untill 28 days
Proportion of patient that received a renal replacement therapy and its duration | 28 days from cannulation
  Number of patient that underwent a renal replacement therapy and duration of renal replacement therapy from cannulation untill 28 days
Duration of vasoactive support | 28 days from cannulation
  Duration of vasoactive drug support from cannulation untill 28 days
Hospital lenght of stay | 28 days from cannulation
  Length of stay from cannulation censored at 90 day
HLA immuno-sensitisation | 28 and 90 days from cannulation
  Proportion of HLA immunosensitisation occuring after cannulation
Proportion of patient with Transfusion related immunologic ( non HLA-related) complications | From randomisation until 28 days
  Transfusion related acute lung injury, hemolytic anemia, irregular antibodies
Proportion of patients with nex onset of sepsis | From randomisation until 28 days
  Sepsis is defined according to Surviving Sepsis Campaign guideline
Proportion of patients with a new onset of acute kidney injury | From randomisation until 28 days
  Acute kidney injury is define according to KDIGO classification
Proportion of patients with liver failure | From randomisation until 28 days
  Liver failure is defined as Hepatic component of SOFA score, Transaminasis Levels
Ischemic stroke | From randomisation until 28 days
  Ischemic stroke is defined as clinical symptoms confirmed by aCT Scan of MRI imaging
Myocardial infarction | From randomisation until 28 days
  According to the Universal definition of myocardial infarction, ESC guidelines
Pulmonary oedema | From randomisation until 28 days
  Dignose by the attending physician based on (Dyspnae, Thoracic X-rays), bowel ischemia ( Abdominal CT or endoscopy proven)
Anaphylactic complications | From randomisation until 28 days
  Anaphylaxis defined according to Ring and Messer Classification
Bowel Ischemia | From randomisation until 28 days
  Proven by Abdominal CT or endoscopy
Cost effectiveness analysis | 28 days, 90 days and 5 years from randomisation
  Actual costs at 28 and 90 days and modelisation for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mouhamed MOUSSA, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service d'Anesthésie-Réanimation CCV Hôpital Cardiologique Centre Hospitalier et Universitaire de Lille, Lille, NORD, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazer CD, Whitlock RP, Fergusson DA, Hall J, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, McGuinness S, Royse A, Carrier FM, Young PJ, Villar JC, Grocott HP, Seeberger MD, Fremes S, Lellouche F, Syed S, Byrne K, Bagshaw SM, Hwang NC, Mehta C, Painter TW, Royse C, Verma S, Hare GMT, Cohen A, Thorpe KE, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Restrictive or Liberal Red-Cell Transfusion for Cardiac Surgery. N Engl J Med. 2017 Nov 30;377(22):2133-2144. doi: 10.1056/NEJMoa1711818. Epub 2017 Nov 12. PMID 29130845
- [Background] Fischer MO, Guinot PG, Debroczi S, Huette P, Beyls C, Babatasi G, Bafi K, Guilbart M, Caus T, Lorne E, Dupont H, Hanouz JL, Diouf M, Abou-Arab O. Individualised or liberal red blood cell transfusion after cardiac surgery: a randomised controlled trial. Br J Anaesth. 2022 Jan;128(1):37-44. doi: 10.1016/j.bja.2021.09.037. Epub 2021 Nov 30. PMID 34862002
- [Result] Vallet B, Robin E, Lebuffe G. Venous oxygen saturation as a physiologic transfusion trigger. Crit Care. 2010;14(2):213. doi: 10.1186/cc8854. Epub 2010 Mar 9. PMID 20236457
- [Result] Aubron C, Cheng AC, Pilcher D, Leong T, Magrin G, Cooper DJ, Scheinkestel C, Pellegrino V. Factors associated with outcomes of patients on extracorporeal membrane oxygenation support: a 5-year cohort study. Crit Care. 2013 Apr 18;17(2):R73. doi: 10.1186/cc12681. PMID 23594433
- [Result] Mazzeffi M, Greenwood J, Tanaka K, Menaker J, Rector R, Herr D, Kon Z, Lee J, Griffith B, Rajagopal K, Pham S. Bleeding, Transfusion, and Mortality on Extracorporeal Life Support: ECLS Working Group on Thrombosis and Hemostasis. Ann Thorac Surg. 2016 Feb;101(2):682-9. doi: 10.1016/j.athoracsur.2015.07.046. Epub 2015 Oct 9. PMID 26443879
- [Result] Holst LB. Benefits and harms of red blood cell transfusions in patients with septic shock in the intensive care unit. Dan Med J. 2016 Feb;63(2):B5209. PMID 26836806
- [Result] Rohde JM, Dimcheff DE, Blumberg N, Saint S, Langa KM, Kuhn L, Hickner A, Rogers MA. Health care-associated infection after red blood cell transfusion: a systematic review and meta-analysis. JAMA. 2014 Apr 2;311(13):1317-26. doi: 10.1001/jama.2014.2726. PMID 24691607
- [Result] Leffell MS, Kim D, Vega RM, Zachary AA, Petersen J, Hart JM, Rossert J, Bradbury BD. Red blood cell transfusions and the risk of allosensitization in patients awaiting primary kidney transplantation. Transplantation. 2014 Mar 15;97(5):525-33. doi: 10.1097/01.tp.0000437435.19980.8f. PMID 24300013
- [Result] Vlaar AP, Hofstra JJ, Determann RM, Veelo DP, Paulus F, Kulik W, Korevaar J, de Mol BA, Koopman MM, Porcelijn L, Binnekade JM, Vroom MB, Schultz MJ, Juffermans NP. The incidence, risk factors, and outcome of transfusion-related acute lung injury in a cohort of cardiac surgery patients: a prospective nested case-control study. Blood. 2011 Apr 21;117(16):4218-25. doi: 10.1182/blood-2010-10-313973. Epub 2011 Feb 16. PMID 21325598
- [Result] Lorusso R, Gelsomino S, Parise O, Mendiratta P, Prodhan P, Rycus P, MacLaren G, Brogan TV, Chen YS, Maessen J, Hou X, Thiagarajan RR. Venoarterial Extracorporeal Membrane Oxygenation for Refractory Cardiogenic Shock in Elderly Patients: Trends in Application and Outcome From the Extracorporeal Life Support Organization (ELSO) Registry. Ann Thorac Surg. 2017 Jul;104(1):62-69. doi: 10.1016/j.athoracsur.2016.10.023. Epub 2017 Jan 26. PMID 28131429
- [Result] Kim HS, Park S. Blood Transfusion Strategies in Patients Undergoing Extracorporeal Membrane Oxygenation. Korean J Crit Care Med. 2017 Feb;32(1):22-28. doi: 10.4266/kjccm.2016.00983. Epub 2017 Feb 28. PMID 31723612
- [Result] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Result] Holst LB, Petersen MW, Haase N, Perner A, Wetterslev J. Restrictive versus liberal transfusion strategy for red blood cell transfusion: systematic review of randomised trials with meta-analysis and trial sequential analysis. BMJ. 2015 Mar 24;350:h1354. doi: 10.1136/bmj.h1354. PMID 25805204
- [Result] Mueller MM, Van Remoortel H, Meybohm P, Aranko K, Aubron C, Burger R, Carson JL, Cichutek K, De Buck E, Devine D, Fergusson D, Follea G, French C, Frey KP, Gammon R, Levy JH, Murphy MF, Ozier Y, Pavenski K, So-Osman C, Tiberghien P, Volmink J, Waters JH, Wood EM, Seifried E; ICC PBM Frankfurt 2018 Group. Patient Blood Management: Recommendations From the 2018 Frankfurt Consensus Conference. JAMA. 2019 Mar 12;321(10):983-997. doi: 10.1001/jama.2019.0554. PMID 30860564
- [Result] Guimbretiere G, Anselmi A, Roisne A, Lelong B, Corbineau H, Langanay T, Flecher E, Verhoye JP. Prognostic impact of blood product transfusion in VA and VV ECMO. Perfusion. 2019 Apr;34(3):246-253. doi: 10.1177/0267659118814690. Epub 2018 Nov 16. PMID 30444173
- [Result] Mazzeffi MA, Tanaka K, Roberts A, Rector R, Menaker J, Kon Z, Deatrick KB, Kaczorowski D, Griffith B, Herr D. Bleeding, Thrombosis, and Transfusion With Two Heparin Anticoagulation Protocols in Venoarterial ECMO Patients. J Cardiothorac Vasc Anesth. 2019 May;33(5):1216-1220. doi: 10.1053/j.jvca.2018.07.045. Epub 2018 Aug 3. PMID 30181084
- [Result] Zeroual N, Blin C, Saour M, David H, Aouinti S, Picot MC, Colson PH, Gaudard P. Restrictive Transfusion Strategy after Cardiac Surgery. Anesthesiology. 2021 Mar 1;134(3):370-380. doi: 10.1097/ALN.0000000000003682. PMID 33475735